CLINICAL TRIAL: NCT02069925
Title: STEP-ED: Reducing Duration of Untreated Psychosis and Its Impact in the U.S.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Harvard University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1310012846; 1R01MH103831-01 (NIH)
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Psychosis; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Detection (ED) (Experimental): This intervention consists of educational campaigns directed at patients & families (who have yet to seek care) and professionals in educational and clinical settings to hasten referral of individuals with new onset psychosis to an established, best-practice first-episode service (i.e. STEP). Interleaved with this educational campaign will be procedures to make the STEP clinic more rapidly responsive to referrals to further shorten the duration of untreated psychosis
  Interventions: Behavioral: Early Detection (ED); Behavioral: Usual Detection
- Usual Detection (Active Comparator): This intervention will provide equivalent best practice care without the benefit of an early detection campaign
  Interventions: Behavioral: Usual Detection

INTERVENTIONS:
Behavioral: Early Detection (ED) — This intervention consists of educational campaigns directed at patients & families (who have yet to seek care) and professionals in educational and clinical settings to hasten referral of individuals with new onset psychosis to an established, best-practice first-episode service (i.e. STEP). Interleaved with this educational campaign will be procedures to make the STEP clinic more rapidly responsive to referrals to further shorten the duration of untreated psychosis
  Arms: Early Detection (ED)
Behavioral: Usual Detection — This intervention will provide equivalent best practice care without the benefit of an early detection campaign

SUMMARY:
The guiding questions for this study are: can a U.S. adaptation of a successful Scandinavian approach (TIPS) to early detection substantially reduce the duration of untreated psychosis (DUP) and improve outcomes beyond an established first-episode service (FES)?

The primary aim of this study is:

1. To determine whether an early detection intervention can reduce DUP in the US, as compared to usual detection. Early detection (ED) will be implemented in one US community (New Haven, CT), and usual detection efforts will continue in another (Boston, MA). DUP will be measured at admission to the corresponding first-episode services (STEP & PREP) in each community, over one year before and throughout ED implementation. The investigators hypothesize that DUP will be reduced significantly in the early detection site compared to the usual detection site;
2. A secondary aim is to determine whether DUP reduction can augment the outcomes of established FES on outcomes in the U.S. The investigators will measure symptoms, functioning and engagement with treatment at entry and over 1 year at each site. The investigators hypothesize that shorter DUP at one FES (STEP) will predict reduced distress and illness severity at entry and better early outcomes at STEP compared to PREP.

DETAILED DESCRIPTION:
Early detection, or reducing the duration of untreated psychosis (DUP) can substantially ameliorate the distress and disability caused by psychotic illnesses. The TIPS project in Scandinavia used a combination of public and targeted education campaigns coupled with rapid availability of comprehensive services to improve the identification, referral and early treatment of psychotic illness. By targeting the dual 'bottlenecks' of inadequate mental health literacy and delayed access to effective treatment, TIPS significantly reduced DUP2 and experimentally demonstrated improved clinical presentations and outcomes.

Effective service models for new onset psychosis exist in the U.S. Multi-element specialty 'first-episode' services (FES), highlighted in this FOA, provide care that is adapted to the specific needs of younger patients and their families and can improve symptoms and functional outcomes during the critical early phase of psychotic illnesses. The NIH-funded Specialized Treatment in Early Psychosis (STEP, New Haven) project, included the first U.S.-based randomized controlled trial to establish the feasibility and effectiveness of a public-sector approach to FES.5 The Prevention and Recovery in Early Psychosis (PREP, Boston) clinic has advanced a similar model of care within an analogous public-academic collaboration.

What is required, as the next logical step, is a test of the effectiveness of TIPS' powerful approach to early detection in a policy-relevant U.S. setting, where relatively fragmented pathways to care raise both the challenges and potential public health impact of early detection. The expertise within the investigators investigative team in the design of early detection and the presence of 2 similar, effective, geographically separated and collaborative FES programs (STEP and PREP) presents an excellent opportunity to conduct such a test and thereby advance secondary prevention for psychotic illnesses in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 35 years old,
* Within first 3 years of psychosis onset (per pre-defined SOS threshold criteria)
* Willing travel to local First Episode Service (STEP, New Haven or PREP, Boston) for treatment;
* Must live in target catchment towns for New Haven site (New Haven, East Haven, West Haven, North Haven, Hamden, Bethany, Orange, Woodbridge, Milford, and Branford) and Boston site (anywhere in Commonwealth of MA)

Exclusion Criteria:

* Established diagnosis of affective psychotic illness (Bipolar disorder or MDD with psychotic features) or psychosis secondary to substance use or a medical illness
* Unable to communicate in English
* IQ<70 or eligible for DDS (Department of Developmental Services) care
* legally mandated to enter treatment or otherwise unable to give free, informed consent
* Unable to reliably determine DUP
* Unstable medical illness

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 285 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Duration of Untreated Psychosis (DUP) | One year before, during campaign and one year after end of campaign
  Time from onset of psychosis to first antipsychotic (DUP-Demand); Time from first antipsychotic to enrollment in STEP/PREP (DUP-Supply); Time from onset of psychosis to enrollment in STEP/PREP (DUP-Total)

SECONDARY OUTCOMES:
Levels of social and occupational functioning | 1 year after enrollment in STEP/PREP
  A trained assessor will administer the positive and negative syndrome scale (PANSS) scale to every subject for levels of social and occupational functioning. The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210.
Change in levels of social and occupational functioning- social | 6 months and 12 months
  The Global Functioning: Social scale will be used, with symptoms rated 1 (most impaired) to 10 (superior functioning).
Change in levels of social and occupational functioning- roles | 6 months and 12 months
  The Global Functioning: Role scale will be used, with symptoms rated 1 (most impaired) to 10 (superior functioning).

OTHER OUTCOMES:
Change in improved labor market / workforce participation and healthcare utilization | 6 months and 12 months
  A trained assessor will administer the Services Utilization and Resources Form for Schizophrenia (SURF) instrument to assess workforce participation and other measures relevant to healthcare utilization. The SURF is a multi-item form that uses participants' or caregivers' report to document comprehensively the number, type, and duration of health services and consumption of non-health resources, such as criminal justice events and public assistance

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Srihari, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Massachusetts Mental Health Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annamalai A, Palmese LB, Chwastiak LA, Srihari VH, Tek C. High rates of obstructive sleep apnea symptoms among patients with schizophrenia. Psychosomatics. 2015 Jan-Feb;56(1):59-66. doi: 10.1016/j.psym.2014.02.009. Epub 2014 Mar 2. PMID 25023923
- [Background] Tek C, Palmese LB, Krystal AD, Srihari VH, DeGeorge PC, Reutenauer EL, Guloksuz S. The impact of eszopiclone on sleep and cognition in patients with schizophrenia and insomnia: a double-blind, randomized, placebo-controlled trial. Schizophr Res. 2014 Dec;160(1-3):180-5. doi: 10.1016/j.schres.2014.10.002. Epub 2014 Oct 29. PMID 25454802
- [Background] Tek C, Kucukgoncu S, Guloksuz S, Woods SW, Srihari VH, Annamalai A. Antipsychotic-induced weight gain in first-episode psychosis patients: a meta-analysis of differential effects of antipsychotic medications. Early Interv Psychiatry. 2016 Jun;10(3):193-202. doi: 10.1111/eip.12251. Epub 2015 May 12. PMID 25962699
- [Background] Kline ER, DeTore NR, Keefe K, Seidman LJ, Srihari VH, Keshavan MS, Guyer M. Development and validation of the client engagement and service use scale: A pilot study. Schizophr Res. 2018 Nov;201:343-346. doi: 10.1016/j.schres.2018.05.006. PMID 29764759
- [Background] Kline E, Thomas L. Cultural factors in first episode psychosis treatment engagement. Schizophr Res. 2018 May;195:74-75. doi: 10.1016/j.schres.2017.08.035. Epub 2017 Aug 30. PMID 28864280
- [Background] van Schalkwyk GI, Davidson L, Srihari V. Too Late and Too Little: Narratives of Treatment Disconnect in Early Psychosis. Psychiatr Q. 2015 Dec;86(4):521-32. doi: 10.1007/s11126-015-9348-4. PMID 25663602
- [Background] Steiner JL, Anez-Nava L, Baranoski M, Cole R, Davidson L, Delphin-Rittmon M, Dike C, DiLeo PJ, Duman RS, Kirk T Jr, Krystal J, Malison RT, Rohrbaugh RM, Sernyak MJ, Srihari V, Styron T, Tebes JK, Woods S, Zonana H, Jacobs SC. The Connecticut Mental Health Center: Celebrating 50 Years of a Successful Partnership Between the State and Yale University. Psychiatr Serv. 2016 Dec 1;67(12):1286-1289. doi: 10.1176/appi.ps.201600373. Epub 2016 Oct 3. PMID 27691379
- [Background] Foss-Feig JH, Adkinson BD, Ji JL, Yang G, Srihari VH, McPartland JC, Krystal JH, Murray JD, Anticevic A. Searching for Cross-Diagnostic Convergence: Neural Mechanisms Governing Excitation and Inhibition Balance in Schizophrenia and Autism Spectrum Disorders. Biol Psychiatry. 2017 May 15;81(10):848-861. doi: 10.1016/j.biopsych.2017.03.005. Epub 2017 Mar 14. PMID 28434615
- [Background] Dixon LB, Goldman HH, Srihari VH, Kane JM. Transforming the Treatment of Schizophrenia in the United States: The RAISE Initiative. Annu Rev Clin Psychol. 2018 May 7;14:237-258. doi: 10.1146/annurev-clinpsy-050817-084934. Epub 2018 Jan 12. PMID 29328779
- [Background] Starc M, Murray JD, Santamauro N, Savic A, Diehl C, Cho YT, Srihari V, Morgan PT, Krystal JH, Wang XJ, Repovs G, Anticevic A. Schizophrenia is associated with a pattern of spatial working memory deficits consistent with cortical disinhibition. Schizophr Res. 2017 Mar;181:107-116. doi: 10.1016/j.schres.2016.10.011. Epub 2016 Oct 10. PMID 27745755
- [Background] Breitborde NJ, Kleinlein P, Srihari VH. Causality Orientations among Individuals with First-Episode Psychosis. Psychosis. 2014 Jun 1;6(2):177-180. doi: 10.1080/17522439.2012.762801. PMID 24976861
- [Background] Hay RA, Roach BJ, Srihari VH, Woods SW, Ford JM, Mathalon DH. Equivalent mismatch negativity deficits across deviant types in early illness schizophrenia-spectrum patients. Biol Psychol. 2015 Feb;105:130-7. doi: 10.1016/j.biopsycho.2015.01.004. Epub 2015 Jan 17. PMID 25603283
- [Background] Guloksuz S, Li F, Tek C, Woods SW, McGlashan TH, Friis S, Srihari VH. Analyzing the Duration of Untreated Psychosis: Quantile Regression. JAMA Psychiatry. 2016 Oct 1;73(10):1094-1095. doi: 10.1001/jamapsychiatry.2016.2013. No abstract available. PMID 27580422
- [Background] Wasser T, Pollard J, Fisk D, Srihari V. First-Episode Psychosis and the Criminal Justice System: Using a Sequential Intercept Framework to Highlight Risks and Opportunities. Psychiatr Serv. 2017 Oct 1;68(10):994-996. doi: 10.1176/appi.ps.201700313. Epub 2017 Sep 1. PMID 28859587
- [Background] Perez VB, Woods SW, Roach BJ, Ford JM, McGlashan TH, Srihari VH, Mathalon DH. Automatic auditory processing deficits in schizophrenia and clinical high-risk patients: forecasting psychosis risk with mismatch negativity. Biol Psychiatry. 2014 Mar 15;75(6):459-69. doi: 10.1016/j.biopsych.2013.07.038. Epub 2013 Sep 16. PMID 24050720
- [Background] Srihari VH, Tek C, Pollard J, Zimmet S, Keat J, Cahill JD, Kucukgoncu S, Walsh BC, Li F, Gueorguieva R, Levine N, Mesholam-Gately RI, Friedman-Yakoobian M, Seidman LJ, Keshavan MS, McGlashan TH, Woods SW. Reducing the duration of untreated psychosis and its impact in the U.S.: the STEP-ED study. BMC Psychiatry. 2014 Dec 4;14:335. doi: 10.1186/s12888-014-0335-3. PMID 25471062
- [Background] Srihari VH, Jani A, Gray M. Early Intervention for Psychotic Disorders: Building Population Health Systems. JAMA Psychiatry. 2016 Feb;73(2):101-2. doi: 10.1001/jamapsychiatry.2015.2821. No abstract available. PMID 26747524
- [Background] Srihari VH. Working toward changing the Duration of Untreated Psychosis (DUP). Schizophr Res. 2018 Mar;193:39-40. doi: 10.1016/j.schres.2017.07.045. Epub 2017 Aug 3. No abstract available. PMID 28779850
- [Background] Mathis WS, Woods S, Srihari V. Blind Spots: Spatial analytics can identify nonrandom geographic variation in first episode psychosis program enrollments. Early Interv Psychiatry. 2018 Dec;12(6):1229-1234. doi: 10.1111/eip.12681. Epub 2018 Jun 21. PMID 29927083
- [Background] Kline E, Hendel V, Friedman-Yakoobian M, Mesholam-Gately RI, Findeisen A, Zimmet S, Wojcik JD, Petryshen TL, Woo TW, Goldstein JM, Shenton ME, Keshavan MS, McCarley RW, Seidman LJ. A comparison of neurocognition and functioning in first episode psychosis populations: do research samples reflect the real world? Soc Psychiatry Psychiatr Epidemiol. 2019 Mar;54(3):291-301. doi: 10.1007/s00127-018-1631-x. Epub 2018 Nov 28. PMID 30488086
- [Derived] Ferrara M, Gallagher K, Yoviene Sykes LA, Markovich P, Li F, Pollard JM, Imetovski S, Cahill J, Guloksuz S, Srihari VH. Reducing Delay From Referral to Admission at a U.S. First-Episode Psychosis Service: A Quality Improvement Initiative. Psychiatr Serv. 2022 Dec 1;73(12):1416-1419. doi: 10.1176/appi.ps.202100374. Epub 2022 Jun 2. PMID 35652190